CLINICAL TRIAL: NCT00446485
Title: Efficacy and Safety of Ginkgo Biloba Standardized Extract (24% Ginkoflavonoglicozides and 6% Terpenes) in Treatment of Mild Cognitive and Concentration Impairment
Brief Title: Efficacy and Safety of Ginkgo Biloba Extract in Mild Cognitive Impairment and Cerebrovascular Insufficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milsing d.o.o. (Other)
Responsible Party: Principal Investigator, Professor of Neurology Vida Demarin, MD, PhD, MD, PhD, FAAN, FAHA, FESO Fellow of Croatian Academy of Sciences and Arts Professor of Neurology, Milsing d.o.o.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MIL-001
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Mild Cognitive Impairment; Cerebrovascular Insufficiency
Keywords: ginkgo biloba; cerebrovascular insufficiency; mild cognitive impairment; concentration impairment
MeSH Terms: conditions — Cognitive Dysfunction; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Ginkgo Biloba standardized extract 24/6
  Interventions: Drug: Ginkgo biloba standardized extract 24/6
- 3 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ginkgo biloba standardized extract 24/6 — tablets, 120 mg/day (60 mg two times daily) during 6 months
  Arms: 1
Drug: Ginkgo Biloba standardized extract 24/6 — tablets, 60 mg/day during 6 months
  Arms: 1
Drug: placebo — placebo during 6 months
  Arms: 3

SUMMARY:
The purpose of the study is to determine weather Ginkgo biloba standardized extract (24% ginkoflavonoglicozides and 6% terpenes) is effective in treatment of cognitive and concentration impairment

DETAILED DESCRIPTION:
Inclusion criteria is cerebrovascular insufficiency MNSE>20. 90 patients are divided into three groups randomly. First group is being administered 120 mg ginkgo biloba extract, second group 60 mg of the extract and the third group has being administered placebo during the period of 6 months. Methods used for evaluation are SCAG, MMSE, MDRS, VFT, CGI, TCD and color Doppler of carotid arteries. Methods used for follow up safety include: routine blood tests, biochemical tests, neurologic and physical examination, vital signs and ECG.

ELIGIBILITY:
Inclusion Criteria:

* cerebrovascular insufficiency and mild cognitive disorder (MMSE=20-28)

Exclusion Criteria:

* pregnancy
* cognitive disorder caused by psychological, metabolic endocrine nutritional and heart disorder
* alcohol or drug abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Changes of MDRS | 6 months
Changes of VFT | 6 months
Changes of CGI | 6 months
Changes of SCAG | 6 months
Changes of MMSE | 6 months

SECONDARY OUTCOMES:
Changes of TCD, and color Doppler of carotid arteries | 6 months
Changes of platelets, hematocrit, prothrombin time, and activated partial tromboplastin time | 6 months
Changes of total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides | 6 months
Safety will be assessed according to occurrence of adverse events during the trial | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vida Demarin, MD PHD, Principal Investigator — University Department of Neurology, Sestre milosrdnice University Hospital, Vinogradska 29, HR-10000 Zagreb, Croatia
Locations (1):
- University Department of Neurology, Sestre milosrdnice University Hospital, Vinogradska 29, Zagreb, Croatia